CLINICAL TRIAL: NCT01162499
Title: Role of Glucagon-Like Peptide-1 in Postprandial Hypoglycemia After Nissen Fundoplication: Studies With the GLP-1 Receptor Antagonist Exendin-(9-39)
Brief Title: Role of Glucagon-Like Peptide-1 in Postprandial Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diva De Leon (Other)
Collaborators: Lester and Liesel Baker Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Diva De Leon, M.D. Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 09-007372
Record Dates: First submitted 2010-05-04; First posted 2010-07-14 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Postprandial Hypoglycemia
Keywords: Post prandial hypoglycemia; hypoglycemia; Nissen fundoplication; Dumping
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39); Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exendin-(9-39) first, then Vehicle (Experimental): After an overnight fast, an intravenous (IV) infusion of Exendin-(9-39) will be started 1 hour prior to the meal challenge and continued for 5 hours. After the first hour of the infusion, subjects will undergo a mixed meal tolerance test in which Pediasure (10cc/kg) will be consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes (for infants under 12 months, Pediasure will be replaced by the infant's formula). Blood samples will be drawn at different time points during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The Exendin-(9-39) dose for the first 3 subjects will be 300pmol/kg/min and, if tolerated, the dose will be increased to 500pmol/kg/min for subsequent subjects.
  The next day, all procedures will be repeated except subjects will receive an IV infusion of normal saline (vehicle) over 6 hours.
  Interventions: Drug: Exendin-(9-39); Other: Vehicle
- Vehicle first, then Exendin-(9-39) (Active Comparator): After an overnight fast, an intravenous (IV) infusion of normal saline (vehicle) will be started 1 hour prior to the meal challenge and continued for 5 hours. After the first hour of the infusion, subjects will undergo a mixed meal tolerance test in which Pediasure (10cc/kg) will be consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes (for infants under 12 months, Pediasure will be replaced by the infant's formula). Blood samples will be drawn at different time points during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1).
  The next day, all procedures will be repeated except subjects will receive an IV infusion of Exendin-(9-39) which will be started 1 hour prior to the meal challenge and continue for 5 hours. The dose for the first 3 subjects will be 300pmol/kg/min and, if tolerated, the dose will be increased to 500pmol/kg/min for subsequent subjects.
  Interventions: Drug: Exendin-(9-39); Other: Vehicle

INTERVENTIONS:
Drug: Exendin-(9-39) — IV infusion of exendin-(9-39) for 5 hours
Other: Vehicle — Normal saline (vehicle) infusion for 5 hours at 0.06 mL/kg/hr
  Other Names: Normal Saline

SUMMARY:
It has been proposed that the rapid gastric emptying of carbohydrate containing fluids into the intestine causes hyperglycemia followed by reactive hypoglycemia. The investigators have shown that glucagon-like peptide-1 (GLP-1) secretion in response to a glucose load is increased in children with Post-prandial hypoglycemia (PPH). This is a proof of concept study to investigate the causative role of GLP-1 in the pathophysiology of PPH after fundoplication by evaluating the effects of GLP-1 receptor antagonism on metabolic variables after a mixed meal.

Hypothesis: In children with post-prandial hypoglycemia after fundoplication, antagonism of the GLP-1 receptor by exendin-(9-39) will elevate nadir blood glucose levels after a meal challenge and prevent post-prandial hypoglycemia.

DETAILED DESCRIPTION:
PPH is a frequent complication of fundoplication in children. The mechanism responsible for the PPH is poorly understood, but involves an exaggerated insulin response to a meal and subsequent hypoglycemia. We have shown that children with PPH after Nissen fundoplication have abnormally exaggerated secretion of GLP-1, an incretin hormone with multiple glucose lowering effects including stimulation of insulin secretion and suppression of glucagon secretion. In this study we seek to examine the causal role of endogenous GLP-1 in PPH after fundoplication by evaluating the effects of antagonizing the GLP-1 receptor with exendin-(9-39) on key metabolic features of PPH.

ELIGIBILITY:
Inclusion Criteria:

* Children (6 months-18 years) who have had fundoplication or other gastric surgeries, irrespective of duration of postoperative period
* Weight > 6.5 Kg
* Signs and/or symptoms of PPH: post-prandial blood glucose levels of < 70 mg/dL ; symptoms including but not limited to feeding difficulties, irritability, nausea, diarrhea, pallor, diaphoresis, weakness, and lethargy after meals

Exclusion Criteria:

* Evidence of a medical condition that might alter results or compromise the elimination of the peptide, including, but not limited to: active infection, kidney failure (creatinine ≥ 2x above upper limit for age), severe liver dysfunction (AST or ALT ≥ 5x upper limit of normal for AST or ALT), severe respiratory or cardiac failure
* Other disorders of glucose regulation such as diabetes mellitus, congenital hyperinsulinism, glycogen storage disease
* Current use (within 1 week) of medications that may alter glucose homeostasis such as glucocorticoids, diazoxide, octreotide
* Use of antihistaminics within 10 days prior to the study
* Moderate and severe anemia defined as a hemoglobin < 10g/dL
* Pregnancy
* Milk and soy protein allergy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diva De Leon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from the Division of Endocrinology and Diabetes at The Children's Hospital of Philadelphia.
Pre-assignment Details: One subject signed consent but they were excluded from study participation after the study team was unable to establish IV access.
Groups:
- Exendin-(9-39) First, Then Vehicle: After an overnight fast, an intravenous (IV) infusion of Exendin-(9-39) was started 1 hour prior to the meal challenge and continued for 4 hours. After the first hour of the infusion, subjects underwent a mixed meal tolerance test in which Pediasure (10cc/kg) was consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes. Blood samples were drawn during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The Exendin-(9-39) dose for the first 3 subjects was 300pmol/kg/min and, as planned, it was increased to 500pmol/kg/min for subsequent subjects. The next day, all procedures were repeated except subjects received an IV infusion of normal saline (vehicle) over 4 hours.
- Vehicle First, Then Exendin-(9-39): After an overnight fast, an intravenous (IV) infusion of normal saline (vehicle) was started 1 hour prior to the meal challenge and continued for 4 hours. After the first hour of the infusion, subjects underwent a mixed meal tolerance test in which Pediasure (10cc/kg) was consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes. Blood samples were drawn to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The next day, all procedures were repeated except subjects received an IV infusion of Exendin-(9-39) which was started 1 hour prior to the meal challenge and continued for 4 hours. The dose for the first 3 subjects was 300pmol/kg/min and, as planned, it was increased to 500pmol/kg/min for subsequent subjects.
Period: Intervention 1 (4 Hours)
Arm/Group | Exendin-(9-39) First, Then Vehicle | Vehicle First, Then Exendin-(9-39)
Started | 3 | 4
Received Intervention | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Unable to establish IV access | 0 | 1
Period: Intervention 2 (4 Hours)
Arm/Group | Exendin-(9-39) First, Then Vehicle | Vehicle First, Then Exendin-(9-39)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all subjects who were randomized and began treatment.
Groups:
- Subject Population: All subjects enrolled and treated in the protocol served as their own control. Because of this and the small sample size, baseline characteristic data is presented together.
Arm/Group | Subject Population
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Previous Surgery [Number; unit: participants]
  Nissen fundoplication | 5
  Gastric pull-through | 1
Feeding Regimen [Number; unit: participants]
  Oral Only | 2
  Both Oral & Gastrostomy | 3
  Gastrostomy Only | 1
Post-Prandial Hypoglycemia Treatment [Number; unit: participants] — Subjects with feeding manipulations had feedings which were modified to decrease volume and slow the rate of delivery.
  participants
    Acarbose | 4
    Feeding | 2
Post-Prandial Hypoglycemia Treatment Frequency [Number; unit: participants]
  Intermittent | 3
  Frequent | 3
Age at Post-Prandial Hypoglycemia Diagnosis [Number; unit: participants]
  Less than 1 year | 1
  Between 1-2 years | 1
  Between 2-3 years | 1
  Between 3-4 years | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Glucose Area Under the Curve (AUC 0-3h)
Description: To examine the effect of Exendin-(9-39) on plasma glucose levels samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (time 0), and then every 30 minutes until 3 hours after the start of the meal. Using this information, the mean plasma glucose area under the curve (AUC) from the start of the infusion to the end of the infusion (3 hours) was calculated for both doses of Exendin-(9-39) [300pmol/kg/min & 500pmol/kg/min] and compared with the vehicle.
Time Frame: 3 hours
Population: Changes were compared between the two dose levels of Exendin-(9-39) of 300pmol/kg/min (3 subjects) and 500pmol/kg/min (3 subjects) were compared to the vehicle infusion (all 6 subjects).
Measure: Mean (Standard Error); unit: mg*min/dl
Groups:
- Exendin-(9-39) 300pmol/kg/Min Dose: After an overnight fast, an intravenous (IV) infusion of Exendin-(9-39) was started 1 hour prior to the meal challenge and continued for 4 hours. After the first hour of the infusion, subjects underwent a mixed meal tolerance test in which Pediasure (10cc/kg) was consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes. Blood samples were drawn during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The Exendin-(9-39) dose was 300pmol/kg/min, infused over 4 total hours.
- Exendin-(9-39) 500pmol/kg/Min Dose: After an overnight fast, an intravenous (IV) infusion of Exendin-(9-39) was started 1 hour prior to the meal challenge and continued for 4 hours. After the first hour of the infusion, subjects underwent a mixed meal tolerance test in which Pediasure (10cc/kg) was consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes. Blood samples were drawn during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The Exendin-(9-39) dose was 500pmol/kg/min, infused over 4 total hours.
- Vehicle: After an overnight fast, an intravenous (IV) infusion of normal saline (vehicle) was started 1 hour prior to the meal challenge and continued for 4 hours. After the first hour of the infusion, subjects underwent a mixed meal tolerance test in which Pediasure (10cc/kg) was consumed by mouth or gastrostomy/nasogastric tube over a period of 15 minutes. Blood samples were drawn during the infusion to measure blood glucose, plasma insulin, glucagon and plasma glucagon-like-peptide-1 (GLP-1). The vehicle was infused over 4 total hours.
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Number analyzed (Participants) | 3 | 3 | 6
mg*min/dl | 22,192.5 (4,784.7) | 25,207.1 (1,157.5) | 21,715.9 (3,597.8)

2. Secondary Outcome: Mean Plasma Insulin Area Under the Curve (AUC 0-3h)
Description: To examine the effect of Exendin-(9-39) on plasma insulin levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (time 0), and then every 30 minutes until 3 hours after the start of the meal. Using this information, the mean plasma insulin area under the curve (AUC) from the start of the infusion to the end of the infusion (3 hours) was calculated for both doses of Exendin-(9-39) [300pmol/kg/min & 500pmol/kg/min] and compared with the vehicle.
Time Frame: 3 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pmol*min/l
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Number analyzed (Participants) | 3 | 3 | 6
pmol*min/l | 14,695.85 (12,662.9) | 9,058.5 (7,562.7) | 19,435.4 (10,392.6)

3. Secondary Outcome: Mean Acetaminophen Plasma Concentration Area Under the Curve (AUC 0-3h)
Description: The effect of gastric emptying was examined using the acetaminophen method whereby acetaminophen (30mg/kg or maximum of 1500mg) was mixed into the Pediasure/formula during the meal tolerance testing. Blood samples were collected every 30 minutes and the absorption of acetaminophen was determined by the gastric emptying rate, as the serum concentrations correlate with gastric emptying of liquids. Mean acetaminophen levels for each group at each time point were used to calculate the Area Under the Concentration versus Time Curve (AUC expressed in μg*min/l) after the consumption of formula for each of the two Exendin-(9-39) dose levels and normal saline vehicle.
Time Frame: 3 hours
Population: AUC were compared between the two dose levels of Exendin-(9-39) of 300pmol/kg/min (3 subjects) and 500pmol/kg/min (3 subjects) were compared to the vehicle infusion (all 6 subjects).
Measure: Mean (Standard Error); unit: μg*min/l
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Number analyzed (Participants) | 3 | 3 | 6
μg*min/l | 3,387.5 (898) | 3,742.8 (124.3) | 3,436.6 (465.2)

4. Secondary Outcome: Peak Plasma Glucagon-like Peptide-1 (GLP-1) Concentration During Infusion
Description: To examine the effect of Exendin-(9-39) on plasma glucagon-like peptide-1 levels, samples were collected at various time points before and during the infusion [Exendin-(9-39) or vehicle] including: 60 minutes before the start of the infusion, again at the start of the infusion (time 0), and then every 30 minutes until 3 hours after the start of the infusion. The mean peak glucagon-like peptide-1 concentration for both Exendin-(9-39) doses were compared with the peak glucagon-like peptide-1 during vehicle infusion.
Time Frame: 60 minutes before the start of the infusion, again at the start of the infusion (time 0), and then every 30 minutes until 3 hours after the start of the infusion
Population: Differences were compared between the two dose levels of Exendin-(9-39) of 300pmol/kg/min (3 subjects) and 500pmol/kg/min (3 subjects) were compared to the vehicle infusion (all 6 subjects).
Measure: Mean (Standard Error); unit: pmol/l
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Number analyzed (Participants) | 3 | 3 | 6
pmol/l | 65.8 (33.3) | 75.2 (5.8) | 72.8 (26.1)

5. Secondary Outcome: Peak Glucagon Concentration During Infusion
Description: To examine the effect of Exendin-(9-39) on plasma glucagon levels, samples were collected at various 3 hours after the start of the infusion. The mean peak glucagon concentration for both Exendin-(9-39) doses were compared with the peak glucagon during vehicle infusion.
Time Frame: as for outcome 4
Population: Differences in peak glucagon concentration were compared between the two dose levels of Exendin-(9-39) of 300pmol/kg/min (3 subjects) and 500pmol/kg/min (3 subjects) were compared to the vehicle infusion (all 6 subjects).
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Number analyzed (Participants) | 3 | 3 | 6
pg/ml | 127.5 (75.7) | 145.7 (33.6) | 114.0 (50.1)

ADVERSE EVENTS:
Time Frame: 30 days following the last administration of study treatment (either Exendin-(9-39) or vehicle)
Arm/Group | Exendin-(9-39) 300pmol/kg/Min Dose | Exendin-(9-39) 500pmol/kg/Min Dose | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exendin-(9-39) 300pmol/kg/Min Dose (N=3) | Exendin-(9-39) 500pmol/kg/Min Dose (N=3) | Vehicle (N=6)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrostomy-tube discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Subject reported discharge from G-tube at home, after completion of study infusions

LIMITATIONS AND CAVEATS:
The primary limitation in addition to small sample size, relates to the fact that none of the subjects experienced significant hypoglycemia during the 3 hour post-meal period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes